CLINICAL TRIAL: NCT03502174
Title: FreeStyle Libre Flash Glucose Monitoring System in Pediatric Populations
Brief Title: FreeStyle Libre Glucose Monitoring System in Pediatric Populations
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-18172
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Subjects will wear the FreeStyle Libre Flash Glucose Monitoring System and will receive no treatment except for safety purposes.

SUMMARY:
This study is a non-randomized, single-arm, multi-center study that is designed to evaluate the safety and effectiveness of the FreeStyle Libre Flash Glucose Monitoring Systems in pediatric populations.

DETAILED DESCRIPTION:
Up to 85 subjects will be enrolled at up to four (4) clinical research sites in the United States. Subjects will wear two Sensors. Each Sensor will have a paired Reader that will be given to the subject. All Readers will be masked during the study (i.e. subjects will not be able to view glucose results obtained from the Sensor on the Reader screen). Subjects will be asked to perform at least 4 capillary Blood Glucose (BG) tests per day using the primary Reader. Interstitial glucose readings from each Sensor will be obtained with the corresponding Readers immediately following each BG test. Subjects will be instructed to report any problems with the device. Subjects will make four (4) to five (5) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Based on the subjects weight, subjects will have up to two (2) in-clinic visits during which intravenous blood draws and YSI reference testing will occur.

ELIGIBILITY:
* Inclusion Criteria:

  * Subject must be at least 6 years of age.
  * Subject must weigh at least 26 kg (57.2 lbs.).
  * Subject must have a diagnosis of type 1 or type 2 diabetes mellitus
  * Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily).
  * Subject must be currently performing at least four (4) capillary blood glucose tests per day.
  * Subject is willing to perform a minimum of 4 finger sticks per day during the study.
  * Subject is willing to allow medical personnel to insert at IV catheter in the arm to allow for venous blood samples to be obtained per the study protocol.
  * Subject and/or guardian must be able to read and understand English.
  * In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
  * Subject must be available to participate in all study visits.
  * Subject must be willing and able to provide written signed and dated informed assent when appropriate.
  * Subject's parent, guardian or legally authorized representative must be willing and able to provide written informed consent.
* Exclusion Criteria:

  * Subject is 18 years of age or older.
  * Subject weighs less than 26 kg (57.2 lbs.).
  * Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
  * Subject is known to be pregnant or becomes pregnant during the study (applicable to female subjects only).
  * Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
  * Subject is currently participating in another clinical trial.
  * Subject has had significant blood loss within 112 days (3.7 months) prior to the beginning of the study activities subjects.
  * Subject is anemic, defined as having hemoglobin levels below 11.5 g/dL for subjects aged 6-11 years old, less than 12.0 g/dL for subjects aged 12-15 years old, less than 12.0 g/dL for females aged 15-17 and less than 13.0 g/dL for males aged 15-171, or as determined by investigator.
  * Subject has X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
  * Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects aged 6-17 years, with type 1 or type 2 diabetes who currently perform capillary blood glucose (BG) testing at least four (4) times a day.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
FreeStyle Libre Flash Glucose Monitoring System Performance | up to 14 days
  System performance will be characterized with respect to YSI reference venous plasma sample measurements. Point accuracy of the system will be evaluated as the proportion of System readings that are within ±20% of the YSI reference value for YSI glucose levels ≥ 80 mg/dl and within ±20 mg/dl for YSI glucose levels <80 mg/dl.
FreeStyle Libre Flash Glucose Monitoring System Related adverse device effects | up to 45 days
  System will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara Alva, PhD, Study Director — Abbot Diabetes care inc.
Locations (3):
- United States (3):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho

IPD SHARING:
Plan to Share IPD: No